CLINICAL TRIAL: NCT00777647
Title: Effect of Carbonated Soft Drinks on Body Weight, Fat Distribution and Metabolic Risk Factors
Brief Title: Effect of Carbonated Soft Drinks on the Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Principal Investigator, Maria Maersk Nielsen, MD, PHD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20070134B
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Metabolic; Complications; Dietary Habits
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Sugar-Sweetened Beverages; Diet, Fat-Restricted; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sugar-sweetened soft drink (Experimental): 54g sugar/L, 180kJ/100mL
  Interventions: Other: Sugar-sweetened soft drink
- Aspartame-sweetened soft drink (Experimental): 1.5kJ/100mL
  Interventions: Other: Aspartame-sweetened soft drink
- Semi-skimmed milk (Active Comparator): 202kJ/100mL
  Interventions: Other: Semi-skimmed milk
- Water (Placebo Comparator): 0kJ/100mL
  Interventions: Other: Water

INTERVENTIONS:
Other: Sugar-sweetened soft drink — One litre a day for six months.
  Arms: Sugar-sweetened soft drink
Other: Aspartame-sweetened soft drink — One litre a day for six months.
  Arms: Aspartame-sweetened soft drink
Other: Semi-skimmed milk — One litre a day for six months
  Arms: Semi-skimmed milk
Other: Water — One litre a day for six months.
  Arms: Water

SUMMARY:
Compared to solid foods, the nutritional energy of drinks may bypass the appetite regulation leading to obesity development. Although drinks sweetened with aspartame are available the anticipated positive effect of these drinks on obesity development has not been convincing. However, the mechanisms linking drinks intake to obesity are yet to be clarified.

The investigators aim is to investigate the long-term effects of intake of soft drinks, milk and water. The study is a parallel, intervention trial with 80 overweight, healthy volunteers. They will be randomly selected to drink one liter a day of one of the four drinks for six months. The objectives are changes in numerous circulating metabolic risk factors, changes in body weight, anthropometric data and fat distribution (measured by DEXA, MRI and MR-spectroscopy).

The investigators expect to clarify the mechanisms linking drinking habits to obesity development and provide scientifically based nutritional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-50 years;
* BMI between 28-36 kg/m2;
* Weight stabile 3 months prior to the study inclusion;
* Less than 10 hours of weekly exercise

Exclusion Criteria:

* Diabetes
* Allergic to phenylalanine or milk
* Smoking
* Pregnancy or breast-feeding

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Body Weight (kg) | Six months
MR spectroscopy | Six months
  to assess liver fat and skeletal muscle fat
Magnetic resonance imaging | Six months
  to assess visceral adipose tissue (VAT) and subcutaneous abdominal adipose tissue (SAAT)
Dual-energy X-ray absorptiometry (DEXA) scan | Six months
  to assess total fat mass (kg), lean body mass (kg), and bone mass (kg)

SECONDARY OUTCOMES:
Blood pressure | Six months
  Systolic and diastolic blood pressure (mmHg)
Circulating metabolic parameters: including serum urate | Six months
  mmol/L
fasting plasma glucose | Six months
  mmol/L
fasting serum insulin | Six months
  pmol/L
Oral Glucose Tolerance Test (OGTT) | Six months
  AUC OGTT glucose and insulin, AUC HOMA-IR, and Matzuda index
Fasting blood lipids | Six months
  Total, LDL, and HDL cholesterol, and TAG (mmol/L)
Fasting plasma FFA | Six months
  mmol/L
Fasting plasma PAI-1 | Six months
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, Professor, Study Chair — Department of Internal Medicine/Endocrinology C, Aarhus University Hospital
Locations (1):
- Department of Internal Medicine/Endocrinology C, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bajahzer MF, Bruun JM, Rosqvist F, Marklund M, Richelsen B, Riserus U. Effects of sugar-sweetened soda on plasma saturated and monounsaturated fatty acids in individuals with obesity: A randomized study. Front Nutr. 2022 Aug 31;9:936828. doi: 10.3389/fnut.2022.936828. eCollection 2022. PMID 36118751
- [Derived] Bruun JM, Maersk M, Belza A, Astrup A, Richelsen B. Consumption of sucrose-sweetened soft drinks increases plasma levels of uric acid in overweight and obese subjects: a 6-month randomised controlled trial. Eur J Clin Nutr. 2015 Aug;69(8):949-53. doi: 10.1038/ejcn.2015.95. Epub 2015 Jun 17. PMID 26081486
- [Derived] Maersk M, Belza A, Stodkilde-Jorgensen H, Ringgaard S, Chabanova E, Thomsen H, Pedersen SB, Astrup A, Richelsen B. Sucrose-sweetened beverages increase fat storage in the liver, muscle, and visceral fat depot: a 6-mo randomized intervention study. Am J Clin Nutr. 2012 Feb;95(2):283-9. doi: 10.3945/ajcn.111.022533. Epub 2011 Dec 28. PMID 22205311